CLINICAL TRIAL: NCT00020124
Title: Phase I and Clinical Pharmacologic Study of Inhaled Doxorubicin in Adults With Advanced Solid Tumors Affecting the Lungs
Brief Title: Inhaled Doxorubicin in Treating Patients With Advanced Solid Tumors Affecting the Lungs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 000088; 00-C-0088; CDR0000067718; NCT00004636 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer; Malignant Mesothelioma; Metastatic Cancer
Keywords: recurrent non-small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; advanced malignant mesothelioma; recurrent malignant mesothelioma; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; pulmonary carcinoid tumor; lung metastases
MeSH Terms: conditions — Lung Neoplasms; Mesothelioma, Malignant; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Doxorubicin

INTERVENTIONS:
Drug: doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving drugs in different ways may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of inhaled doxorubicin in treating patients who have advanced solid tumors affecting the lungs.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and phase II dose of inhaled doxorubicin in patients with advanced solid tumors affecting the lungs.
* Determine the toxicity of this regimen in these patients.
* Determine the pharmacokinetic profile of inhaled doxorubicin in blood in these patients.
* Determine the relationship between pharmacodynamic parameters and toxic effects of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive inhaled doxorubicin every 3 weeks for up to 3 doses. Patients with stable or responding disease may receive additional doses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of doxorubicin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 3 weeks and 3 months.

PROJECTED ACCRUAL: Approximately 33 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven advanced cancer not curable by standard chemotherapy, radiotherapy, or surgery

  * Clinical evidence of primary lung or tracheal cancer OR
  * Metastatic cancer to the lung
* Extrathoracic metastases eligible if following criteria are met:

  * Sites are stable
  * Pulmonary sites are primary life-threatening sites
  * Evidence that study treatment may benefit the patient
* Measurable or evaluable disease
* No germ cell tumor, leukemia, or lymphoma involving the lungs that is treatable with systemic agents
* No complete atelectasis due to high-grade airway obstruction

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* More than 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 1.0 mg/dL
* AST and ALT less than 1.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.6 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* LVEF at least 40% by MUGA scan or echocardiogram
* No unstable angina, congestive heart failure, or symptomatic arrhythmias

Pulmonary:

* DLCO at least 50% predicted
* FVC and FEV1 at least 50% predicted
* Resting oxygen saturation at least 90%
* Exercise oxygen saturation at least 85%
* Oxygen consumption greater than 50% predicted
* No prior radiation pneumonitis
* No asthma
* No radiation-induced pulmonary damage

Other:

* No hypersensitivity to doxorubicin
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study
* HIV negative
* No congenital problems (e.g., cleft palate) or other anomalies that prevent tight fit of a mouthseal

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy and recovered
* No prior trastuzumab (Herceptin)

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and recovered
* Prior doxorubicin allowed if LVEF at least 40% by MUGA scan or echocardiogram
* No prior mitomycin, bleomycin, or nitrosoureas
* No other concurrent systemic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* At least 12 months since prior radiotherapy to chest
* No prior radiotherapy to more than 20% of total lung volume
* Prior chest wall or primary breast radiotherapy allowed
* Prior radioactive iodine allowed
* No concurrent thoracic radiotherapy

Surgery:

* See Disease Characteristics
* No prior total pneumonectomy

Other:

* No other concurrent experimental drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Schrump, MD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States